CLINICAL TRIAL: NCT06483490
Title: Mitochondrial Dysfunction and Immune Checkpoints in Chronic Obstructive Pulmonary Disease (COPD) and Lung Cancer: the Role of Environmental Pollutants
Brief Title: Environmental Pollutants in COPD and Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Cardarelli Hospital (Other)
Responsible Party: Principal Investigator, Prof. Bruno D'Agostino, PhD, MD, Prof, University of Campania Luigi Vanvitelli
Other Study IDs: MITO2024
Record Dates: First submitted 2024-06-19; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: COPD and Lung Cancer
Keywords: COPD; Lung cancer; Mitochondrial dysfunction; immune checkpoints; Environmental pollution; cross-sectional; non-pharmacological; multicenter study
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Neoplasms; Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biopsies, bronco-alveolar lavage (BAL) and blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is a cross-sectional, non pharmacological study — Measurement of immune checkpoint levels, mitochondrial dysfunction, pollutant concentrations and G-quadruplex levels and their correlation in all enrolled subjects.

SUMMARY:
Epidemiological studies describe a statistically significant correlation between hospitalization rate and exposure to environmental pollutants such as atmospheric particulates (PM10 and PM2.5) and polycyclic aromatic hydrocarbons (PAH). Indeed, they induced the release of inflammation mediators and oxidative stress, involved in remodeling and destruction of the alveolar parenchyma, in turn associated with the respiratory disease onset and progression such as asthma, COPD, pulmonary fibrosis and lung cancer. Interestingly, oxidative stress associated with environmental pollutants could also induce DNA damage by affecting the stability of G-quadruplex (G4) sequences. Given the role of G4 in physiological and pathological processes and their presence in mitochondrial DNA, telomeres and proto-oncogene promoters, it is interesting to investigate the potential involvement in cellular mechanisms of response to oxidative stress associated with pollutants. Moreover, it is known that pollutant-induced oxidative stress has the ability to alter mitochondrial integrity, leading to mitochondrial dysfunction. The mitochondria involvement in the innate and adaptive immune response regulation corroborates the role of pollutants in respiratory diseases pathogenesis. Indeed, mitochondrial function and integrity are critical for both the effector and memory stages of differentiation of T cells which play a primary role in respiratory diseases. In this context, the PD-1/PD-L1 immune check-points are essential in promoting the immune system homeostasis. Currently, although the role of environmental pollutants, mitochondrial dysfunction and the PD-1/PD-L1 axis in the pathogenesis of many respiratory diseases is recognized, it is useful to further clarify the underlying molecular interconnections and the mechanisms by which pollutants could affect mitochondrial integrity and immune checkpoints.

DETAILED DESCRIPTION:
Epidemiological studies describe a statistically significant correlation between hospitalization rate and exposure to environmental pollutants such as atmospheric particulates (PM10 and PM2.5). The harmfulness to human health depends on both the chemical composition and the particle size. Chronic exposure to particulate matter contributes to the risk of developing respiratory and cardiovascular diseases as well as may increase the risk of lung cancer. In fact, particulate matter is universally recognized as a Class 1 carcinogen. The fine particulates are harmful for human health by the ability to carry other pollutants such as polycyclic aromatic hydrocarbons (PAHs) to the lungs. Notably, the PAHs cause lung damage due to their ability to induce the release of inflammatory mediators and oxidative stress. These events result in remodeling and destruction of the alveolar parenchyma, both involved in respiratory disease onset and progression such as asthma, COPD, pulmonary fibrosis, and lung cancer. Therefore, the involvement of environmental pollutants in the predisposition and exacerbation of lung diseases, in the development of respiratory infections and in the process of carcinogenesis is evident. Moreover, in addition, oxidative stress associated with environmental pollutants could induce DNA damage. Recently, unconventional DNA structures have been identified, recognized as G-quadruplex (G4), which are particularly susceptible to oxidative stress. In fact, it is known that guanine-rich DNA sequences are more reactive with hydroxyl radicals than guanine residues scattered throughout the genome, and that oxidative damage (8-oxo-dg) formation at the G4 level reduces its thermal stability. Given the role of G4 in physiological and pathological processes and their presence in mitochondrial DNA, telomeres and proto-promoters oncogenes, it is interesting to investigate the potential involvement in cellular mechanisms of response to oxidative stress associated with pollutants. It is known that pollutant-induced oxidative stress has the ability to alter mitochondrial integrity, leading to mitochondrial dysfunction. Recent evidence points to innate immunity, apoptosis, and metabolism being largely regulated by mitochondrial activities. In turn, normal mitochondrial activity can be affected by inflammatory processes, infections, tobacco smoking and "environmental insults" and could respond to such stimuli through structural alterations and protein expression resulting in dysfunction. The mitochondria involvement in the innate and adaptive immune response regulation corroborates the role of pollutants in respiratory diseases pathogenesis. Indeed, mitochondrial function and integrity are critical for both the effector and memory stages of differentiation of T cells which play a primary role in respiratory diseases. In this context, the PD-1/PD-L1 immune check-points are essential in promoting the immune system homeostasis. Indeed, they take part in self-tolerance and consist of a series of ligand-receptor interactions involved in coordinating an effective immune response while limiting collateral damage to organs and tissues. The contribution of our research group in the study of the pathway PD-1/PD-L1 in the context of respiratory diseases was relevant, observing that this pathway is not only altered in lung cancer but also in chronic lung diseases such as COPD. Currently, although the role of environmental pollutants, mitochondrial dysfunction and the PD-1/PD-L1 axis in the pathogenesis of many respiratory diseases is recognized, it is useful to further clarify the underlying molecular interconnections and the mechanisms by which pollutants could affect mitochondrial integrity and immune checkpoints.

ELIGIBILITY:
Inclusion Criteria:

* All patients of both sexes and over the age of 18 years
* Clinical diagnosis of suspected lung cancer

Exclusion Criteria:

* Patients with infectious diseases,
* Patients with interstitiopathy
* Patients with autoimmune diseases
* Patients with cancers not covered by the inclusion criteria
* subjects on glucocorticoid therapy
* subjects who cannot undergo bronchial biopsy
* subjects who will not sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients belong to UOC Interventional Pulmonology- Hospital Cardarelli and subjected to bronchoscopy, BAL and routine blood sampling following the clinical routine. All participants must sign the informed consent for participation in the study. All analyses to be carried out in this study will not require more human samples than is required by normal clinical practice. The excess amount of biological samples will be destroyed.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Immune checkpoints in COPD and lung cancer. | The outcome will be measured once for each included patient after the enrollment through study completion, an average of 3 year
  Measurement of immune checkpoint PD-L1, PD-1, e CTLA-4 levels in all enrolled subjects. The relative expression will be calculated by Real-time PCR using the comparative cycle threshold method (Ct) (2 - ΔΔCt).
Mitochondrial activity in COPD and lung cancer. | The outcome will be measured once for each included patient after the enrollment through study completion, an average of 3 year.
  Measurement of mitochondrial dysfunction markers in all enrolled subjects. ATP levels will be measured by means of the 'ATP bioluminescence assay kit' and the factors 'PTEN-induced kinase 1 (PINK)-Parkin-mediated pathway' (marker of mitophagy) and sirtuins (marker of senescence) by ELISA assay
Environmental pollutants in COPD and lung cancer. | The outcome will be measured once for each included patient after the enrollment through study completion, an average of 3 year.
  Measurement of pollutant concentrations in all enrolled subjects. A fraction of BAL and peripheral blood will be used for the analysis of pollutants deposited on the cell surface and in the supernatant by means of gas chromatography (GC) coupled to mass spectrometry (MS).
G-quadruplex levels in all enrolled subjects. | The outcome will be measured once for each included patient after the enrollment through study completion, an average of 3 year.
  Measurement of G-quadruplex levels in all enrolled subjects. The BG4 antibody will be used to evaluate the formation of G-quadruplex structures. Laser scanning confocal microscopy will be performed with a laser scanning confocal microscope with a 400X objective and the signal analysed with Fiji software.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardarelli Hospital, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilkinson TMA. Immune checkpoints in chronic obstructive pulmonary disease. Eur Respir Rev. 2017 Jun 28;26(144):170045. doi: 10.1183/16000617.0045-2017. Print 2017 Jun 30. PMID 28659497
- [Background] Durham AL, Adcock IM. The relationship between COPD and lung cancer. Lung Cancer. 2015 Nov;90(2):121-7. doi: 10.1016/j.lungcan.2015.08.017. Epub 2015 Aug 29. PMID 26363803
- [Background] Wasen C, Erlandsson MC, Bossios A, Ekerljung L, Malmhall C, Toyra Silfversward S, Pullerits R, Lundback B, Bokarewa MI. Smoking Is Associated With Low Levels of Soluble PD-L1 in Rheumatoid Arthritis. Front Immunol. 2018 Jul 27;9:1677. doi: 10.3389/fimmu.2018.01677. eCollection 2018. PMID 30140263
- [Background] Prakash YS, Pabelick CM, Sieck GC. Mitochondrial Dysfunction in Airway Disease. Chest. 2017 Sep;152(3):618-626. doi: 10.1016/j.chest.2017.03.020. Epub 2017 Mar 21. PMID 28336486
- [Background] Sachdeva K, Do DC, Zhang Y, Hu X, Chen J, Gao P. Environmental Exposures and Asthma Development: Autophagy, Mitophagy, and Cellular Senescence. Front Immunol. 2019 Nov 29;10:2787. doi: 10.3389/fimmu.2019.02787. eCollection 2019. PMID 31849968